CLINICAL TRIAL: NCT04436900
Title: Evaluation of Macular Structural and Functional Function Following Extensive Retinal Laser Therapy in Patients With Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1396.455
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 20 patients (40 eyes) with PDR underwent PRP with ARC with a spot number of 1,200 to 1,500 per eye and spot size 500 micron with a duration of 200 ms.
  Interventions: Procedure: Panretinal Photocoagulation (PRP)

INTERVENTIONS:
Procedure: Panretinal Photocoagulation (PRP) — PRP with ARC with a spot number of 1,200 to 1,500 per eye and spot size 500 micron with a duration of 200 ms.

SUMMARY:
The present study is a semi-experimental clinical trial that 20 patients (40 eyes) with PDR underwent PRP with ARC with a spot number of 1,200 to 1,500 per eye and spot size 500 micron with a duration of 200 ms. The variables of contrast sensitivity, macula thickness under fovea , BCVA, the width of thyroid under fovea , RNFL thickness in the four areas around the disc, and the quality of life questionnaire of all patients were recorded at the beginning of the study.Retinal and choroid under fovea thickness and RNFL thickness were assessed in four areas, one week and one month after the end of treatment, and all the variables mentioned earlier were evaluated three months after PRP surgery.

This study is single group that the outcomes are compared before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2 with PDR
* Having conscious satisfaction

Exclusion Criteria:

* Patients with a history of other eye diseases
* Patients with a history of previous laser treatment
* Patients with a history of injection of Anti-VGEF
* Patients with Vitreous hemorrhage
* Patients with Macula edema
* Patients with myopia more than -3 diopters or hyperopiamore than +3 diopters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Life Quality | up to 3 months
  A generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral, social environment as well as health and disease Which is measured by a quality of life questionnaire
RNFL | up to 30 days
  retinal nerve fiber layer which measured by PP-OCT (optical coherence tomography)
BCVA | up to 3 months
  best corrected visual acuity which measured by SD-OCT
Retinal thickness in the central part of Fovea | up to 30 days
  Measured by SD-OCT
Choroid thickness in the central part of Fovea | up to 30 days
  Measured by EDI-OCT
Physical examination of PDR | up to 3 months
  An eye exam performed by an ophthalmologist will determine if there is retinopathy
Contrast sensitivity | up to 3 months
  Contrast sensitivity which measured by Melbourne edge test
Angiography with fluorescein | up to 3 months
  By injecting fluorescein into the vein and then taking an X-ray to diagnose PDR

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran